CLINICAL TRIAL: NCT07170527
Title: Long-Term Outcomes and Post-Intensive Care Syndrome: An Explorative, Prospective, Observational Cohort Study to Investigate the Associations Between Metabolic Signatures and Physical Functioning in Critically Ill Patients
Brief Title: Long-Term Outcomes and Post-Intensive Care Syndrome: Investigating the Associations Between Metabolic Signatures and Physical Functioning in Critically Ill Patients
Acronym: TOPICS
Status: Recruiting | Type: Observational
Sponsor: ARH van Zanten, MD PhD (Other)
Collaborators: Danone Global Research & Innovation Center (Industry); Wageningen University and Research (Other); TKI Agri & Food (Unknown)
Responsible Party: Sponsor-Investigator, ARH van Zanten, MD PhD, Principal investigator, Gelderse Vallei Hospital
Organization: Gelderse Vallei Hospital (Other)
Other Study IDs: NL87540.091.24
Record Dates: First submitted 2025-08-30; First posted 2025-09-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Post-Intensive Care Syndrome (PICS)
Keywords: Post-Intensive Care Syndrome (PICS); Critical illness; Intensive Care Unit (ICU); Recovery; Long-Term Outcomes
MeSH Terms: conditions — postintensive care syndrome; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Adult patients with an expected ICU length of stay of ≥72 hours, or who receive (non-) invasive mechanical ventilation (IMV or NIV) within 48 hours after ICU admission with an expected ventilatory support duration of at least 48 hours.

SUMMARY:
Despite being young, healthy, and physically fit, some intensive care unit (ICU) patients experience significantly worse functional recovery after critical illness than older patients with multiple comorbidities although a poor precondition seems to be associated with worse ICU outcomes. This paradox highlights a fundamental gap in our understanding of the determinants of long-term recovery. While nonmodifiable factors such as age and pre-existing disease explain part of the variation, they cannot fully account for the wide heterogeneity in outcomes. Metabolic disturbances during critical illness, such as hypercatabolism, impaired muscle metabolism, nutritional deficits, systemic inflammation, and disruption of gut health, are likely to influence recovery trajectories, yet remain poorly characterized. Because these processes represent potentially modifiable targets, combining their evaluation with nonmodifiable patient characteristics is essential for unraveling the complex, multifactorial mechanisms underlying post-intensive care syndrome (PICS).

This explorative, prospective, observational study aims to investigate the associations between metabolic signatures during the acute phase of critical illness and PICS outcomes throughout the recovery trajectory of ICU survivors, with a primary focus on physical functioning. In addition, the study explores the longitudinal course of metabolic parameters from ICU admission up to 12 months post-discharge, and whether these signatures can help identify distinct recovery phenotypes.

Participants will be followed for 12 months, with study assessments at ICU admission, ICU discharge, and at 3-, 6-, and 12-months post-ICU admission.

DETAILED DESCRIPTION:
Yearly, more than 70.000 patients are admitted to the intensive care unit (ICU) in the Netherlands. Although survival rates from critical illness have improved over the last decades, still patients suffer from profound weakness and functional impairments, collectively referred to as post-intensive care syndrome (PICS). PICS encompasses a cluster of long-lasting physical, cognitive, and mental health problems that have a severe impact on patients' quality of life. Studies investigating strategies to improve recovery after critical illness have shown limited effectiveness. This might be due to heterogeneous recovery trajectories observed among ICU survivors. Research has focussed on the associations between non-modifiable factors (e.g., age, sex and disease severity) and PICS outcomes. However, comprehensive assessment of potentially modifiable metabolic signatures (such as hypercatabolism, muscle metabolism, nutritional status, inflammatory response, and gut health) is lacking. These modifiable factors might be of interest as these likely shape the recovery trajectory of critical illness survivors. This approach, by combining the assessment of nonmodifiable factors together with potentially modifiable factors, is essential for understandiing the complex, multifactorial, pathophysiological mechanisms underlying PICS.

The TOPICS study aims to explore the associations between modifiable factors during critical illness (such as hypercatabolism, muscle metabolism, nutritional status, inflammatory response, and gut health), and physical and psychological functioning in ICU survivors. The main questions it aims to answer are:

1. What are the associations between metabolic signatures during the acute phase of critical illness and physical functioning 3-months post-ICU admission?
2. What are the associations between metabolic signatures during the acute phase of critical illness and physical functioning across different time points in the recovery phase?
3. What are the associations between metabolic signatures during the acute phase of critical illness and psychological functioning (cognitive functioning and mental health status) across different time points during the recovery phase?
4. What is the trajectory of PICS outcomes, quality of life and metabolic parameters during one year following ICU admission?
5. Can distinct patient phenotypes with different recovery trajectories be identified based on metabolic and physical functioning outcomes?

The study is a monocentre, longitudinal, explorative, prospective, observational study. Study measurements will be performed upon ICU admission, and in the recovery period (ICU discharge, 3-, 6-, and 12-months post-ICU admission). Study procedures include:

1. Completion of questionnaires on health-related quality of life, cognitive functioning, mental health status, and sleep quality.
2. Assessment of physical functioning.
3. Collection of blood samples.
4. Collection of fecal samples.
5. Assessment of dietary intake.

The study population will consist of 200 adult patients admitted to the ICU of Gelderse Vallei Hospital, Ede, who receive (non-) invasive mechanical ventilation (IMV or NIV) within 48 hours after ICU admission and are expected to receive ventilatory support for at least 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of ICU admission;
* Received ventilatory support (IMV or NIV) within 48 hours after ICU admission with an expected duration of ≥48 hours during ICU stay (irrespective of ICU length of stay); OR
* An expected ICU length of stay of ≥72 hours (irrespective of ventilatory support).

Exclusion Criteria:

* Concurrent participation in an intervention study with an anticipated therapeutic effect on PICS outcomes (physical functioning, cognitive functioning, or mental health status)
* Pre-admission diagnosis of a progressive neurological disease (e.g., Alzheimer's disease, Parkinson's disease, amyotrophic lateral sclerosis, progressive forms of multiple sclerosis)
* Participants with neurological paralysis significantly affecting leg function (e.g., spinal cord injury, multiple sclerosis)
* Patients receiving palliative care, with a life expectancy of <3 months (e.g., hospice care or equivalent)
* Patients who are moribund (i.e., in the final stages of a terminal illness, with imminent death expected)
* Anticipated logistical limitations during recovery phase (e.g., transfer to another hospital, no fixed abode);
* Deemed not suitable to participate based upon the judgement of the treating intensivist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 200 adult patients admitted to the ICU of Gelderse Vallei Hospital, Ede, with an expected ICU length of stay of ≥72 hours, or who receive invasive mechanical ventilation (IMV) or non-invasive ventilation (NIV) within 48 hours after ICU admission and are expected to receive this ventilatory support (IMV or NIV) for ≥48 hours.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Subjective physical functioning | 3-months post-ICU admission
  Assessed by the Physical Component Score (PCS) of the Short Form-36 (SF-36) questionnaire, ranging from 0 to 100. Scores above or below the average of 50 indicate better or worse physical health compared to the general population, respectively.
Handgrip strength | 3-months post-ICU admission
  Assessed with Jamar dynamometer, measured in kilograms (kg).
Leg strength and endurance | 3-months post-ICU admission
  Assessed by the 30-second chair stand test (30sCST)
Muscle size | 3-months post-ICU admission
  Assessed by muscle ultrasound of the quadriceps muscles
Muscle size | 3-months post-ICU admission
  Assessed by calf circumference, measured in cm
Body composition | 3-months post-ICU admission
  Assessed by bio-electrical impedance analysis (BIA)

SECONDARY OUTCOMES:
Subjective physical functioning | 3 times during cohort (at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed by the Physical Component Score (PCS) of the Short Form-36 (SF-36) questionnaire, ranging from 0 to 100. Scores above or below the average of 50 indicate better or worse physical health compared to the general population, respectively.
Handgrip strength | 3 times during cohort (at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed with Jamar dynamometer, measured in kilograms (kg)
Leg strength and endurance | 3 times during cohort (at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed by the 30sCST
Muscle size | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed by muscle ultrasound of the quadriceps muscles
Muscle size | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed by calf circumference, measured in cm
Body composition | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 6- and 12-months post-ICU admission)
  Assessed by BIA
Cognition | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Abbreviated 14-item Cognitive Failure Questionnaire (CFQ-14), ranging from 0 to 56. A higher score indicates more cognitive errors.
Cognition | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Montreal Cognitive Assessment (MoCA), ranging from 0 to 30. A higher score indicates better cognition.
Anxiety | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Hospital Anxiety and Depression Scale (HADS), ranging from 0 to 42. Questions 1, 3, 5, 7, 9, 11 and 13 measure symptoms of anxiety (range: 0-21). Higher scores indicate worse symptoms of anxiety.
Depression | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Hospital Anxiety and Depression Scale (HADS), ranging from 0 to 42. Questions 2, 4, 6, 8, 10, 12 and 14 measure symptoms of depression (range: 0-21). Higher scores indicate worse symptoms of depression.
Post-traumatic stress disorder | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Trauma Screening Questionnaire (TSQ), ranging from 0 to 10. A higher score indicates worse symptoms of Post-Traumatic Stress Disorder.
Health-related Quality of Life | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Short Form 36 (SF-36), ranging from 0 to 100. A higher score indicates a better Health-related Quality of Life.
Sleep quality | 4 times during cohort (at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Pittsburgh Sleep Quality Index (PSQI), ranging from 0 to 21. Higher scores indicate worse sleep quality.
Level of independence | 4 times during cohort (ICU admission, 3-, 6- and 12-months post-ICU admission)
  Barthel index, ranging from 0-20. Higher scores indicate higher independence of the participant.
Frailty | 5 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, 6- and 12-months post-ICU admission)
  Rockwood Clinical Frailty Scale (CFS), ranging from 1 to 9. A higher score indicates a more severe degree of frailty.
Dietary intake | 2 times during cohort (3-, and 12-months post-ICU admission)
  24-hour recall, combined with a dietary food record.
Lipid metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma triglycerides, total cholesterol, HDL-cholesterol, and LDL-cholesterol levels
Glucose metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma glucose levels
Glucose metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma insulin levels
Glucose metabolism | 3 times during cohort (at ICU admission, 3-, and 12-months post-ICU admission)
  Blood HbA1c levels
Protein metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma amino acid levels
Thyroid hormones | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma thyroid hormone levels
Markers for kidney function | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma kidney function markers
Markers for liver function | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma liver function markers
Markers for muscle metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma muscle metabolism markers
Micronutrient levels | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Blood micronutrient levels
Systemic inflammation markers | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma systemic inflammation marker levels
Neuro-inflammation markers | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma neuro-inflammation marker levels
Intestinal inflammation markers | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Fecal intestinal inflammation marker levels
Microbiota composition | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Microbiota composition in feces (e.g., abundance, diversity and function)
Intestinal fermentation markers | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Fecal fermentation marker levels
Intestinal integrity markers | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Serum and plasma intestinal integrity marker levels
Short-chain fatty acids (SCFA) and branched-chain fatty acids (BCFA) | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma and fecal SCFA and BCFA concentrations
Tryptophan metabolism | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Plasma tryptophan metabolite levels
Haematological health | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Mean corpuscular volume
Haematological health | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Haemoglobin levels
Haematological health | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Haematocrit levels
Haematological health | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Leucocyte levels
Haematological health | 4 times during cohort (at ICU admission, at ICU discharge (an average of 10 days), 3-, and 12-months post-ICU admission)
  Thrombocyte levels

CONTACTS AND LOCATIONS:
Locations (1):
- Gelderse Vallei Hospital, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared upon reasonable request.